CLINICAL TRIAL: NCT00252837
Title: A 24-Week Randomized, Double-Blind, Parallel-Group, Multi-Centre, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Tesaglitazar Therapy When Administered as Monotherapy to Drug-Naïve Patients With Type 2 Diabetes
Brief Title: GALLANT 22 Tesaglitazar vs. Placebo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00055; EudraCT No 2004-004374-90
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar; Diet

INTERVENTIONS:
Drug: Tesaglitazar
Behavioral: Dietary and Lifestyle counseling

SUMMARY:
This is a 24-week randomized, double-blind, parallel-group, multi-center, placebo-controlled study of tesaglitazar (0.5 and 1 mg) in patients with type 2 diabetes, not adequately controlled on diet and lifestyle advice alone during the run-in period. The study comprises a 6-week single-blind placebo run-in period, followed by 24-week treatment period and a 3-week follow-up period.

The study design of GALLANT 2 is identical to GALLANT 22; the blinded study data from GALLANT 2 will be transferred to the GALLANT 22 database and will be analyzed together with the data from GALLANT 22 clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents
* Drug-naïve (ie, no use of antidiabetic drug[s], for at least 24 weeks prior to visit 1).

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475
Dates: Start 2005-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to end of randomized treatment period in glycosylated hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Changes in the following variables from baseline to the end of the randomized treatment period:
Lipid parameters (triglyceride [TG], total cholesterol, high-density lipoprotein cholesterol [HDL C], non-HDL C, low-density lipoprotein cholesterol [LDL C], apolipoproteins [Apo] A-I, Apo B, Apo CIII, free fatty acids, lipoprotein particle size and c
C-reactive protein, LDL C/HDL C ratio and Apo B/Apo A-I ratio
Fasting plasma glucose (FPG), homeostasis assessment model, insulin, proinsulin, C-peptide
Tumor necrosis factor-alpha, intracellular adhesion molecule-1
Fibrinogen
Proportion of patients with microalbuminuria
Waist/hip ratio
Responder analyses for HbA1c, FPG, TG, HDL C, non HDL C and LDL C according to pre-specified values
Proportion of patients reaching pre-specified target levels for HbA1c, FPG, TG, HDL C, non-HDL C and LDL C
Pharmacokinetics of tesaglitazar
Safety and tolerability of tesaglitazar by assessment of adverse events, laboratory values, electrocardiogram,, pulse, blood pressure, hypoglycemic events, body weight, cardiac evaluation, and physical examination
Patient-reported outcomes: Well-Being Questionnaire (W BQ12)
Audit of Diabetes Dependent Quality of Life (ADDQoL). ADDQoL will only be applied in Poland.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (101):
- Australia (9):
  - Research Site, Adelaide
  - Research Site, Cairns
  - Research Site, Gosford
  - Research Site, Keswick
  - Research Site, Kippa-Ring
  - Research Site, Melbourne
  - Research Site, Miranda
  - Research Site, Nowra
  - Research Site, Wollongong
- Czechia (9):
  - Research Site, Brno
  - Research Site, Hodonín
  - Research Site, Hradec Králové
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Semily
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
- Estonia (5):
  - Research Site, Paide
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
  - Research Site, Viljandi
- France (7):
  - Research Site, Angers
  - Research Site, Briollay
  - Research Site, Poitiers
  - Research Site, Saint-Benoît
  - Research Site, Saint-Ouen
  - Research Site, Toulouse
  - Research Site, Trélazé
- Greece (2):
  - Research Site, Athens
  - Research Site, Piraeus
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Székesfehérvár
- Latvia (7):
  - Research Site, Daugavpils
  - Research Site, Jēkabpils
  - Research Site, Madona
  - Research Site, Riga
  - Research Site, Sigulda
  - Research Site, Talsi
  - Research Site, Valmiera
- Lithuania (4):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Panevezys
  - Research Site, Vilnius
- Norway (11):
  - Research Site, Aursmoen
  - Research Site, Bergen
  - Research Site, Enebakk
  - Research Site, Fredrikstad
  - Research Site, Haugesund
  - Research Site, Hønefoss
  - Research Site, Inderøy
  - Research Site, Larvik
  - Research Site, Lierskogen
  - Research Site, Oslo
  - Research Site, Rolvsøy
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (19):
  - Research Site, Katowice, Ochojec
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Radom
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Toruñ
  - Research Site, Tychy
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zielona Góra
- Research Site, Belgrade, Serbia and Montenegro
- Slovakia (10):
  - Research Site, Dolný Kubín
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Ľubochňa
  - Research Site, Nové Zámky
  - Research Site, Považská Bystrica
  - Research Site, Šahy
  - Research Site, Trenčín
  - Research Site, Veľký Meder
  - Research Site, Žilina
- Sweden (9):
  - Research Site, Åmål
  - Research Site, Borås
  - Research Site, Gothenburg
  - Research Site, Mölndal
  - Research Site, Partille
  - Research Site, Skene
  - Research Site, Stenungsund
  - Research Site, Uddevalla
  - Research Site, Vänersborg